CLINICAL TRIAL: NCT03751488
Title: A Randomized, Single-Dose, Open-Label, Parallel-Group Study to Determine the Relative Pharmacokinetic Characteristics of LY03010 Versus INVEGA SUSTENNA® in Schizophrenia Patients
Brief Title: A Study to Determine Pharmacokinetic Characteristics of LY03010 Versus INVEGA SUSTENNA® in Schizophrenia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY03010/CT-USA-101
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2018-12

CONDITIONS: Schizo Affective Disorder; Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY03010 351mg (Experimental): LY03010 at 351 mg
  Interventions: Drug: LY03010
- LY03010 156 mg (Experimental): LY03010 at 156 mg
  Interventions: Drug: LY03010
- LY03010 117mg (Experimental): LY03010 at 117mg
  Interventions: Drug: LY03010
- INVEGA SUSTENNA (Active Comparator): INVEGA SUSTENNA 156mg
  Interventions: Drug: Invega Sustenna 156 MG in 1 ML Prefilled Syringe

INTERVENTIONS:
Drug: LY03010 — Single Dose of LY03010 at 351 mg or 156 mg or 117mg
  Arms: LY03010 117mg; LY03010 156 mg; LY03010 351mg
Drug: Invega Sustenna 156 MG in 1 ML Prefilled Syringe — Single Dose at 156mg
  Arms: INVEGA SUSTENNA

SUMMARY:
This study will look at the Characteristics of LY03010 Versus INVEGA SUSTENNA® in the blood of Schizophrenia Patients

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent and complying with study procedures;
2. Have an identified support person (e.g., family member, case worker, social worker) considered reliable by the Investigator to help ensure compliance with study visits and to alert staff of any issues of concern;
3. Have a stable place of residence for the 3 months prior to screening and throughout the study;
4. Male or female ≥18 to ≤65 years of age who meets diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-V) for at least 1 year before screening;
5. Be on a stable dose of oral antipsychotic medication(s) other than risperidone, paliperidone, clozapine, ziprasidone, or thioridazine for at least 4 weeks prior to screening;
6. Be clinically stable based on clinical assessments and a Positive and Negative Syndrome Scale (PANSS) total score ≤70 as well as a PANSS HATE (hostility, anxiety, tension and excitement) subtotal score <16 at screening;
7. Clinical Global Impression-Severity (CGI-S) score of 1 to 4, inclusive;
8. Body mass index (BMI) ≥17.0 and ≤37 kg/m2; body weight ≥50 kg;
9. Creatinine level within the normal range;
10. All female patients (childbearing potential and non-childbearing potential) must have a negative pregnancy test result at both screening and baseline. Female patients must meet 1 of the following 3 conditions: (i) postmenopausal for at least 12 months without an alternative medical cause, (ii) surgically sterile (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal occlusion) based on patient report, or (iii) if of childbearing potential (WOCBP), practicing or agree to practice a highly effective contraception method of birth control. Highly effective methods of birth control include an intrauterine device (IUD), intrauterine hormone-releasing system (IUS), and contraceptives (oral, skin patches, or implanted or injectable products) using combined or progestogen-only hormonal contraception associated with inhibition of ovulation. A vasectomized male partner is an acceptable birth control method if the vasectomized partner is the sole sexual partner of the female patient and the vasectomized partner has received medical confirmation of surgical success. Highly effective methods of birth control must be used for at least 14 days prior to study drug dosing, throughout the study, and for another 80 days after the end-of-treatment (EOT) visit (or at least 200 days after the dose, whichever is longer) to minimize the risk of pregnancy;
11. Sexually active fertile male patients must be willing to use acceptable contraception methods (such as double barrier methods of a combination of male condom with either cap, diaphragm or sponge with spermicide) from study drug dosing, throughout the study, and for another 80 days after the EOT visit (or at least 200 days after the dose, whichever is longer) if their partners are women of childbearing potential.

Exclusion Criteria:

1. Primary and active DSM-V Axis I diagnosis other than schizophrenia or schizoaffective disorder;
2. Patients who meet DSM-V criteria for substance abuse (moderate or severe) with the exception of caffeine or nicotine in the past 6 months prior to screening, or test positive for a drug of abuse or alcohol at screening or baseline (except positive findings that can be accounted for by documented prescriptions used as prescribed by a treating physician as a part of the treatment for the patient's psychiatric illness);
3. History of treatment resistance, defined as failure to respond to 2 adequate treatment regimens (minimum of 4 weeks at the patient's maximum tolerated dose) of different antipsychotic medications;
4. Known or suspected hypersensitivity or intolerance of risperidone, paliperidone, or any of their excipients (oral risperidone tolerability test will be completed during the screening period, approximately 14 days prior to dosing, for patients without documented evidence [medical record or written statement from a licensed medical practitioner who has treated the patient] of tolerating risperidone or paliperidone, and patients who show an allergic reaction to this test will be excluded from the study);
5. Known non-responders to risperidone or paliperidone;
6. Patients who pose a significant risk of a suicide attempt based on history or the Investigator's judgment; answer "yes" to Suicidal Ideation items 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) for current or past 30 days on the "Baseline/Screening version" at screening; have had suicidal behavior in the last 12 months as measured by the C-SSRS at screening; or are at imminent risk of suicide or violent behavior based on the Investigator's clinical assessment or the C-SSRS assessment of lifetime suicidal ideation or behavior at screening;
7. Any one or more of the following 3 conditions: (i) clinically significant liver dysfunction, (ii) hepatitis B surface antigen (HBsAg) positive, or (iii) a serum alanine transaminase (ALT) or aspartate transaminase (AST) > 2x upper limit of normal (ULN) range (if the ALT or AST levels are between 2x and 3x ULN in the first screening test and the elevation may be caused by non-specific reasons in the judgment of the Investigator, a second test can be performed after one week. If the repeated ALT or AST levels are still >2x ULN, the patient must not be included in the study). However, patients who are hepatitis C positive may be enrolled, if this condition is considered stable without treatment and liver function is normal;
8. History of symptomatic orthostatic hypotension with a decrease of ≥20 mmHg in systolic blood pressure (SBP) or decrease of ≥10 mmHg in diastolic blood pressure (DBP) when changing from supine to standing position after having been in the supine position for at least 5 minutes or SBP less than 105 mmHg in a supine position at screening;
9. Uncontrolled diabetes or hemoglobin A1c (HbAlc) level ≥7%, or newly diagnosed within the past 12 months prior to screening;
10. History of neuroleptic malignant syndrome (NMS) or tardive dyskinesia; history of severe akathisia or extra-pyramidal reactions such as dystonia with previous use of risperidone or other neuroleptic treatments; score ≥ 3 on the Global Clinical Assessment of the BARS; or score ≥ 1 on the AIMS at screening. Patients who experience mild extrapyramidal symptoms attributable to study medications will be allowed to continue with appropriate anticholinergic treatment (benztropine, diphenhydramine, and/or trihexyphenidyl);
11. Electroconvulsive therapy within 60 days before screening;
12. Use of a long-acting injectable for the treatment of schizophrenia within 4 weeks (8 weeks for Risperdal Consta®) before screening;
13. Use of injectable paliperidone palmitate within 10 months before screening;
14. Use of clozapine within 4 weeks before screening;
15. Use of nonselective or irreversible monoamine oxidase inhibitor (MAOI) antidepressants within 30 days before screening;
16. Use of other antidepressants unless the patient has been on a stable dose for at least 30 days before screening;
17. Use of strong inducers of either CYP 3A4 or P-glycoprotein (P-gp) within 2 weeks or 5 half-lives, whichever is longer, before screening;
18. QTcF interval greater than 450 msec for males and 470 msec for females or a prior history or presence of circumstances that could increase the risk of torsade de pointes or sudden death in association with the use of drugs that prolong the QTc interval, or other clinically significant ECG findings in the opinion of the Investigator;
19. Clinically significant past medical history (within 2 years) of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, renal, hepatic, bronchopulmonary, neurologic, immunologic disorders, or drug hypersensitivity which, in the judgement of the Investigator, would interfere with the patient's ability to participate in the study;
20. Malignancies with the exception of basal cell or squamous cell skin cancer or in situ cervical cancer within 5 years prior to screening;
21. History or current diagnosis of epilepsy or convulsive disorder other than a single childhood febrile seizure;
22. Participation in a previous clinical study of paliperidone or any other related medications within the past 3 months prior to screening;
23. Receipt of another investigational product within 1 month, or 5 half-lives of the other investigational product, whichever is longer, prior to screening;
24. Donation or blood collection of > 1 unit (approximate 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to screening;
25. Any clinical observation or clinical laboratory abnormality including human immunodeficiency virus (HIV) positive test result or abnormal ECG findings at screening or baseline visits which, in the opinion of the Investigator, may endanger the patient or interfere with the endpoints of the study. If the results of clinical laboratory or ECG testing are outside normal reference ranges, the patient may be enrolled but only if these findings are determined not to be clinically significant by the Investigator. This determination must be recorded in the patient's source documents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
AUC | Time Zero to Last quantifiable concentration (120 days)
  Area under the concentration
CMax | 120 days
  Maximum observed concentration
Tmax | 120 days
  Time to Reach Cmax

SECONDARY OUTCOMES:
Safety Assessments as measured by Adverse Events that occur during the study | 120 days
  Safety Assessments as measured by Adverse Events that occur during the study

CONTACTS AND LOCATIONS:
Overall Officials: Amy Sun, MD PhD, Study Director — Luye Pharma
Locations (2):
- United States (2):
  - Collaborative Neuroscience Network LLC, Garden Grove, California
  - Hassman Research Institute, Berlin, New Jersey

IPD SHARING:
Plan to Share IPD: No